CLINICAL TRIAL: NCT00164138
Title: Development of an Intervention and and Education Program for Adult Women With Urinary Incontinence and Chronic Lung Disease Including Cystic Fibrosis (CF) and Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Prevalence and Treatment of Urinary Incontinence in Women With Cystic Fibrosis and Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108/01; Dept. of Health and Aged Care
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Incontinence; physiotherapy; treatment; pelvic floor muscle function; coughing; forced expirations; lung disease
MeSH Terms: conditions — Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive; Cough; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pelvic Floor Training Group (Experimental): Pelvic floor training, biofeedback.
  Interventions: Procedure: Pelvic floor training group

INTERVENTIONS:
Procedure: Pelvic floor training group — pelvic floor training, electrotherapy, bladder retraining.

SUMMARY:
Women with chronic lung disease characterised by chronic cough report urinary incontinence. Recently there have been reports of increased urinary incontinence in girls and women with cystic fibrosis. While coughing is a known risk factor for stress incontinence, other risk factors and causes are poorly understood in this population. Treatment of incontinence for patients with chronic lung disease is also poorly addressed, adding to the burden of disease for women with chronic lung disease, carers and the health system. This project will estimate the prevalence of women with CF and COPD compared to healthy age matched controls and will evaluate the effect of a specific treatment and management program for these patients. The results will be disseminated to respiratory health professionals. We hypothesise that women with chronic cough will have a higher incidence of urinary incontinence than healthy controls and that a specific treatment program will result in alleviation of the problems and improved quality of life.

DETAILED DESCRIPTION:
This project will be undertaken in two phases:

Phase 1 will involve a mailed out screening questionnaire survey of a sample of 50-60 women with CF and 50-60 women with COPD to investigate the prevalence of incontinence in these populations. For subjects requiring assistance an independent physiotherapist is available to assist them with completion of the questionnaire over the telephone. Return stamped addressed envelopes will be provided to each subject in the initial mail-out. The following types of incontinence will be investigated: stress incontinence, urge incontinence, faecal incontinence, faecal urgency, nocturnal enuresis, voiding dysfunction, insensible urine loss, defaecation difficulty, known prolapse, childhood enuresis.

Phase 2 will be an assessment and interventional study. Subjects will be measured before and after the treatment intervention and followed up for three months using the following validated outcome measures:

* Symptoms measures: 3-day frequency-volume chart, 24-hour pad weigh test, 7-day accident diary, quality of life measure (King's Health Questionnaire).
* Pelvic floor muscle function:

  * Electromyographic study (EMG) of the pelvic floor muscles using an intravaginal electrode
  * Transabdominal diagnostic ultrasound
* Adherence to program: self report diary.

Subjects being assessed for pelvic floor muscle activity will attend the School of Physiotherapy Movement Laboratory to undertake the following tests:

1. A 7-day accident diary
2. King's Health Questionnaire
3. Severity index score
4. ICIQ SF score
5. Ultra-sound examination of movement of the pelvic floor muscles
6. EMG measurement of pelvic floor muscle activity.

Ultrasound measurement using an Acoustic Imaging Performa ultrasound unit (Dornier, Medtech, USA) and its accompanying software will be used for imaging and measurement. The aim is to obtain images showing the greatest degree of displacement during pelvic floor muscle activity. The mean value of three recorded measurement will be used for statistical analysis for the following activities: 20 second maximum effort endurance hold, 3 deep coughs, 3 huffs.

EMG pelvic floor activity will be measured using an intravaginal electrode at rest, following a brief maximum voluntary contraction over 1 second and a sustained maximum voluntary contraction over 20 seconds to determine the strength and timing of pelvic floor muscle activity in subjects with chronic cough compared to healthy controls. In order to investigate pelvic floor muscle activity during forced expirations and coughing EMG recording will be recorded with thoracic movement during huffing and coughs and during the preceding inspiration.

The effects of a physiotherapeutic intervention over a three-month period on incontinence will be investigated. All subjects will be referred for treatment to one of 9 selected continence physiotherapists working in continence clinics or women's health practices providing state of the art treatment conveniently located for each subject. Treatment will comprise standard physiotherapy interventions with up to 5 treatments within the 3-months period customised on the basis of the assessment. Details of treatments will subsequently be examined for broad consistency. Pelvic floor muscle training, biofeedback, electrotherapy and bladder training will be included in treatment as individually indicated.. A further assessment will occur immediately post-treatment program followed by a follow-up assessment 3-months after the completion of the treatment program. Results of the study will be provided to medical practitioners and physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* Women with CF and COPD

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2001-12; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Symptom measures:
3-day frequency volume chart,
24 hour pad weigh test,
accident diary,
quality of life using King's Health Questionnaire.
pelvic floor muscle function:
Trans-abdominal diagnostic ultra-sound
EMG study of the pelvic floor muscles

CONTACTS AND LOCATIONS:
Overall Officials: Brenda M Button, DPhty, PhD, Principal Investigator — The Alfred; John W Wilson, MBBS, PhD, Study Director — The Alfred
Locations (2):
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - School of Physiotherapy, The University of Melbourne, Melbourne, Victoria